CLINICAL TRIAL: NCT02432144
Title: A Long-Term Open-Label Treatment and Extension Study of UX003 rhGUS Enzyme Replacement Therapy in Subjects With MPS 7
Brief Title: A Study of UX003 Recombinant Human Beta-Glucuronidase (rhGUS) Enzyme Replacement Therapy in Subjects With Mucopolysaccharidosis Type 7, Sly Syndrome (MPS 7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX003-CL202; 2015-001875-32 (EudraCT Number)
Expanded Access: NCT03775174 (Available)
Record Dates: First submitted 2015-04-22; First posted 2015-05-01 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Sly Syndrome; MPS VII; Mucopolysaccharidosis; Mucopolysaccharidosis VII
Keywords: MPS 7; Sly Syndrome; MPS VII; Enzyme Replacement Therapy; Rare Disease; Mucopolysaccharidosis Type 7; Lysosomal Storage Disease; Metabolic Disorder
MeSH Terms: conditions — Mucopolysaccharidosis VII; Mucopolysaccharidoses; Rare Diseases; Lysosomal Storage Diseases; Metabolic Diseases | interventions — vestronidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UX003 (Experimental): 4 mg/kg UX003 every other week (QOW)
  Interventions: Drug: UX003

INTERVENTIONS:
Drug: UX003 — solution for intravenous (IV) infusion
  Other Names: recombinant human beta-glucoronidase; rhGUS; Mepsevii ™; vestronidase alfa; vestronidase alfa-vjbk

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of UX003 in subjects with MPS 7.

DETAILED DESCRIPTION:
Participants with MPS 7 who were UX003 treatment-naïve or previously enrolled and treated in a prior clinical study of UX003 (e.g. UX003-CL301 [NCT02230566], investigator sponsored trials, expanded access/compassionate use) can enroll into this treatment and extension study provided all eligibility criteria is met for a given participant.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPS 7 based on leukocyte or fibroblast glucuronidase enzyme assay or genetic testing.
* Willing and able to provide written, signed informed consent or, in the case of subjects under the age of 18 (or 16 years, depending on the region), provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Willing and able to comply with all study procedures.
* Sexually active subjects must be willing to use acceptable, highly-effective methods of contraception while participating in the study and for 30 days following the last dose.
* Females of childbearing potential must have a negative pregnancy test at Baseline and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have not experienced menarche, or have had tubal ligation at least one year prior to completion of the primary study, or have had total hysterectomy.
* For UX003 treatment-naïve subjects only, apparent clinical signs of lysosomal storage disease as judged by the Investigator, including at least one of the following: enlarged liver and spleen, joint limitations, airway obstruction or pulmonary problems, limitation of mobility while still ambulatory.
* For UX003 treatment-naïve subjects only, elevated urinary glycosaminoglycans (uGAG) excretion at a minimum of 2-fold over normal.
* For UX003 treatment-naïve subjects only, aged 5 years and older.

Exclusion Criteria:

* If enrolled in a prior UX003 clinical study, the subject experienced safety-related event(s) in the prior UX003 clinical study that, in the opinion of the Investigator and sponsor, precludes resuming UX003 treatment.
* Undergone a successful bone marrow or stem cell transplant or has any degree of detectable chimaerism with donor cells.
* Presence or history of any hypersensitivity to rhGUS or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects.
* Pregnant or breastfeeding at Baseline or planning to become pregnant (self or partner) at any time during the study.
* Other than the use of UX003, use of any investigational product (drug or device or combination) within 30 days prior to Baseline, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Presence of a condition of such severity and acuity that, in the opinion of the Investigator, warrants immediate surgical intervention or other treatment or may not allow safe study participation.
* Concurrent disease or condition, or laboratory abnormality that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or introduce additional safety concerns.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals, Inc.
Locations (7):
- United States (4):
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of Minnesota, Minneapolis, Minnesota
  - Baylor College of Medicine, Houston, Texas
- Hospital Infantil Candido Fontoura Sao Paulo, São Paulo, Brazil
- Centenario Hospital Miguel Hidalgo, Pediatrics, Aguascalientes, Mexico
- Unidade de Doenças Metabólicas - Centro Hospitalar do Porto, Porto, Portugal

REFERENCES:
- [Result] Wang RY, da Silva Franco JF, Lopez-Valdez J, Martins E, Sutton VR, Whitley CB, Zhang L, Cimms T, Marsden D, Jurecka A, Harmatz P. The long-term safety and efficacy of vestronidase alfa, rhGUS enzyme replacement therapy, in subjects with mucopolysaccharidosis VII. Mol Genet Metab. 2020 Mar;129(3):219-227. doi: 10.1016/j.ymgme.2020.01.003. Epub 2020 Jan 11. PMID 32063397
- [Derived] Montano AM, Rozdzynska-Swiatkowska A, Jurecka A, Ramirez AN, Zhang L, Marsden D, Wang RY, Harmatz P. Growth patterns in patients with mucopolysaccharidosis VII. Mol Genet Metab Rep. 2023 Jun 26;36:100987. doi: 10.1016/j.ymgmr.2023.100987. eCollection 2023 Sep. PMID 37415957
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with mucopolysaccharidosis VII (MPS 7) who were UX003 treatment-naïve or previously enrolled and treated in a prior clinical study of UX003 could enroll into this treatment and extension study provided all eligibility criteria had been met for a given participant.
Pre-assignment Details: Ten of 12 participants entered this extension study at study Week 0 with ongoing UX003 treatment for the prior 24 or 48 weeks in study UX003-CL301 [NCT02230566]; 2 participants had a large gap between studies (61 weeks between doses).
Period: Overall Study
Arm/Group | UX003
Started | 12
Completed (Includes 8 participants who switched to commercially available vestronidase alfa before Week 144.) | 11
Not Completed | 1
Not completed — Participant Non-Compliance | 1

BASELINE CHARACTERISTICS:
Groups:
- UX003: 4 mg/kg UX003 QOW
Arm/Group | UX003
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.56 (5.466)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9
  Other, Not Specified | 3
Urinary Glycosaminoglycans (uGAG) [Mean (Standard Deviation); unit: g GAG/g creatinine] | 1.54848 (0.413237)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: An adverse event (AE) is defined as any untoward medical occurrence, whether or not considered drug related. A serious AE is an AE that at any dose, results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect; or is an important medical event. AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), Grade 5 (death). TEAEs were defined as reported AEs with onset during the treatment.
Time Frame: From first dose of study drug until 30 days after the last dose of study drug. Mean duration of UX003 treatment was 100.5 weeks.
Population: Full Analysis Set: all enrolled participants who received at least one dose of investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | UX003
Number analyzed (Participants) | 12
Participants
  TEAEs | 12
  Serious TEAEs | 4
  Treatment-Related TEAEs | 9
  Treatment-Related Serious TEAEs | 1
  Grade 3 or 4 TEAEs | 3
  TEAEs Leading to Treatment Discontinuation | 0
  TEAEs Leading to Study Discontinuation | 0
  TEAEs Leading to Death | 0

2. Secondary Outcome: Percent Change From Baseline Over Time in Urinary Glycosaminoglycan (uGAG) Excretion (Liquid Chromatography-Tandem Mass Spectrometry, Dermatan Sulfate)
Description: First morning void urine was evaluated for uGAG concentration and normalized to urinary creatinine concentration.
Time Frame: Baseline (prior to the first dose of study drug in UX003-CL301), Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Full Analysis Set: all enrolled participants who received at least one dose of investigational product in this study; participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage change in uGAG excretion
Arm/Group | UX003
Number analyzed (Participants) | 12
percentage change in uGAG excretion
  Week 0 | -62.19 (16.133)
  Week 12: number analyzed (Participants) | 11
  Week 12 | -67.31 (13.953)
  Week 24 | -64.03 (14.669)
  Week 36: number analyzed (Participants) | 11
  Week 36 | -60.58 (23.552)
  Week 48: number analyzed (Participants) | 10
  Week 48 | -57.04 (23.611)
  Week 60: number analyzed (Participants) | 9
  Week 60 | -72.25 (18.609)
  Week 72: number analyzed (Participants) | 9
  Week 72 | -78.52 (10.367)
  Week 84: number analyzed (Participants) | 8
  Week 84 | -80.89 (10.023)
  Week 96: number analyzed (Participants) | 8
  Week 96 | -82.39 (6.011)
  Week 108: number analyzed (Participants) | 7
  Week 108 | -82.19 (6.551)
  Week 120: number analyzed (Participants) | 5
  Week 120 | -88.74 (4.023)
  Week 132: number analyzed (Participants) | 4
  Week 132 | -89.22 (3.662)
  Week 144: number analyzed (Participants) | 4
  Week 144 | -91.62 (1.827)
Statistical Analysis 1: Comparison: UX003; Week 0; Test type: Superiority; p < 0.0001, GEE model — P-values are from generalized estimating equation (GEE) model including baseline value and visit (in this study) as a categorical variable. The covariance structure within subjects is assumed to be exchangeable; LS Mean = -62.28, 95% CI 2-sided [-71.98 to -52.59], Standard Error of Mean 4.946
Statistical Analysis 2: Comparison: UX003; Week 12; Test type: Superiority; p < 0.0001, GEE model — P-values are from a GEE model including baseline value and visit (in this study) as a categorical variable. The covariance structure within subjects is assumed to be exchangeable; LS Mean = -67.18, 95% CI 2-sided [-73.49 to -60.86], Standard Error of Mean 3.224
Statistical Analysis 3: Comparison: UX003; Week 24; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 2, analysis 2]; LS Mean = -64.12, 95% CI 2-sided [-71.99 to -56.24], Standard Error of Mean 4.016
Statistical Analysis 4: Comparison: UX003; Week 36; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 2, analysis 2]; LS Mean = -60.80, 95% CI 2-sided [-72.54 to -49.06], Standard Error of Mean 5.992
Statistical Analysis 5: Comparison: UX003; Week 48; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 2, analysis 2]; LS Mean = -57.85, 95% CI 2-sided [-71.87 to -43.82]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after the last dose of study drug. Mean duration of UX003 treatment was 100.5 weeks.
Description: TEAEs, defined as reported AEs with onset during the treatment, are presented.
Arm/Group | UX003
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UX003 (N=12)
Gastroenteritis (Infections and infestations) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UX003 (N=12)
Eosinophilia (Blood and lymphatic system disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 2
Otorrhoea (Ear and labyrinth disorders) | 1
Conjunctivitis Allergic (Eye disorders) | 2
Eye Pruritus (Eye disorders) | 1
Lacrimation Increased (Eye disorders) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3
Gingival Bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Lip Ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 1
Tooth Discolouration (Gastrointestinal disorders) | 1
Tooth Loss (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chest Pain (General disorders) | 1
Fatigue (General disorders) | 1
Gait Disturbance (General disorders) | 1
Infusion Site Extravasation (General disorders) | 5
Infusion Site Swelling (General disorders) | 2
Oedema Peripheral (General disorders) | 2
Pyrexia (General disorders) | 2
Seasonal Allergy (Immune system disorders) | 1
Abscess Neck (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Otitis Externa (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Otitis Media Acute (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 3
Root Canal Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Tinea Pedis (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 7
Viral Infection (Infections and infestations) | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 2
Skin Abrasion (Injury, poisoning and procedural complications) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal Instability (Musculoskeletal and connective tissue disorders) | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain Compression (Nervous system disorders) | 1
Cervical Cord Compression (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hydrocephalus (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Memory Impairment (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sensory Disturbance (Nervous system disorders) | 1
Sinus Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Somnambulism (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 2
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02432144/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT02432144/SAP_001.pdf